CLINICAL TRIAL: NCT07040202
Title: Evaluating Immune Responses to Dengue and Sepsis in Hospitalized Patients in Cambodia
Brief Title: Immune Responses to Dengue and Sepsis
Acronym: DEN-SEP
Status: Recruiting | Type: Observational
Sponsor: Institut Pasteur du Cambodge (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 092 NECHR; Approval number (Other: National Ethics Committee for Health Research Cambodia)
Record Dates: First submitted 2025-05-25; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Dengue; Sepsis
Keywords: dengue; sepsis; observational; infection
MeSH Terms: conditions — Dengue; Sepsis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy controls: Participants with no chronic illness, no regular medications, no febrile illness in 28 days, no diagnosis of or treatment for dengue or bacterial infection in the past 6 months.
- Patients with dengue-like illness: Patients presenting with dengue-like symptoms for a duration of maximum 72h before inclusion. Dengue-like symptoms include: presentation with oral temperature >38°C AND at least two of the following symptoms suggestive of dengue-like illness: headache, retro-orbital pain, myalgia, joint pain, rash, any bleeding symptoms, nausea or vomiting, lethargy or restlessness, abdominal pain, liver enlargement.
- Sepsis patients: Patients admitted for less than 48 hours with a primary diagnosis of sepsis as per treating team AND have blood cultures ordered AND on empiric antibiotics due to concern for bacterial infection.

SUMMARY:
The goal of this research study is to help the investigators better understand serious dengue disease. The investigators will collect clinical information and up to four blood samples from participants with dengue, sepsis, or healthy people. The investigators will perform multiple analyses on the blood samples and compare results between dengue patients and those with sepsis and healthy people.

DETAILED DESCRIPTION:
This is an observational study enrolling n=200 hospitalized individuals with dengue-like illness, n=30 individuals with sepsis, and n=10 healthy controls to evaluate immune responses in plasma leak syndromes. Sepsis and dengue patients will have blood collected at enrollment, day 1, and day 3, and dengue patients will have an additional blood draw at day 21. Healthy participants will have a single blood draw at enrollment. The blood collected will enable the evaluation of immune kinetics, including changes in neutrophils, cytokines, and adaptive responses, as dengue progresses or improves. Overall, this study will facilitate the evaluation of an understudied cell type and will provide unique data for understanding the temporal changes in the immune response to dengue virus. A better understanding of dengue pathophysiology will help identify potential therapeutic targets to improve outcomes in this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dengue-like illness:

Patients presenting with dengue-like symptoms for a duration of maximum 72h before inclusion. Dengue-like symptoms include: presentation with oral temperature >38°C AND at least two of the following symptoms suggestive of dengue-like illness: headache, retro-orbital pain, myalgia, joint pain, rash, any bleeding symptoms, nausea or vomiting, lethargy or restlessness , abdominal pain, liver enlargement

* Sepsis patients:

Patients admitted for less than 48 hours with a primary diagnosis of sepsis as per treating team AND have blood cultures ordered AND on empiric antibiotics due to concern for bacterial infection.

* Healthy controls:

Participants with no chronic illness, no regular medications, no febrile illness in 28 days, no diagnosis of or treatment for dengue or bacterial infection in the past 6 months.

Exclusion Criteria:

* For biobanking purposes, children less than 2 years of age, and individuals who are pregnant, pregnant within the last 90 days, and/or breastfeeding are excluded due to restrictions on the blood volumes and the repeated sampling times.
* Individuals that do not provide informed consent will not be included for the study.
* Severe/chronic/recurrent pathological conditions: clinically significant autoimmune disease or immunodeficiency (including history of organ transplant), haematologic disorders, cardiac diseases, diabetes, cancer, HIV, chronic hepatic or renal insufficiency.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within the 6 months prior to the inclusion. For corticosteroids, this will mean a dose equivalent to 20 mg/day of prednisone or equivalent for > 2 weeks (inhaled and topical steroids allowed)
* Chronic administration of NSAIDs, including aspirin: prolonged intake (>2 weeks) within 6 months before study or any intake within the 7 days preceding sampling [exception for low dose aspirin: maximum 250mg/daily]
* Any underlying, chronic, or current condition that, in the opinion of the investigator, may interfere with their participation in the study.
* Expected death in the next 48-hours

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be enrolled from Kampong Speu District Referral Hospital (Kampong Speu), Preah Kossamak Hospital (Phnom Penh), and the International Center of Excellence in Research Cambodia.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of low density neutrophils in mild/moderate vs severe dengue | From enrollment to study day 3
  Low density neutrophils will be isolated from the PBMC layer of centrifuged blood and characterized via flow cytometry. The percentages of low density neutrophils will be compared between dengue groups.
Mean florescence intensity of neutrophils expressing spleen tyrosine kinase | From enrollment to study day 3.
  The mean florescence intensity (MFI) of neutrophils expressing spleen tyrosine kinase will be measured via flow cytometry and compared between mild/moderate vs severe dengue.
Serum level of myeloperoxidase in mild/moderate versus severe dengue. | Enrollment to study day 3
  The serum level of myeloperoxidase will be measured in pg/mL and compared between participants with mild/moderate versus severe dengue.

SECONDARY OUTCOMES:
Percentage of low density neutrophils in dengue versus sepsis | From enrollment to study day 3
  Low density neutrophils will be isolated from the PBMC layer of centrifuged blood and characterized via flow cytometry. The percentage of low density neutrophils will be compared in dengue versus sepsis.
Mean florescence intensity of neutrophils expressing spleen tyrosine kinase in dengue versus sepsis | From enrollment to study day 3.
  Mean florescence intensity (MFI) of neutrophils expressing spleen tyrosine kinase will be measured via flow cytometry and compared between those with dengue versus sepsis. Other markers of neutrophil maturation, activation, and degranulation will be measured by flow cytometry and compared among dengue groups and between dengue and sepsis.
Serum level of myeloperoxidase in dengue versus sepsis | Enrollment to study day 3
  Serum level of myeloperoxidase will be measured in pg/mL and compared between participants with dengue versus sepsis. Other biomarkers of neutrophil activation such as calprotectin, resistin, and lactoferrin will be measured and compared among groups.
Serum levels of interferon-gamma and interleukin-10 (pg/mL) | Enrollment through day 3.
  Serum levels of interferon-gamma and interleukin-10 (pg/mL) will be measured and compared between dengue groups and sepsis overtime. Other cytokines may also be measured and compared among groups.
Percentage of DENV-specific activated T cells | Enrollment through day 21.
  Activation induced marker assays will be used to compare dengue virus (DENV)-specific T cell activation over time in mild/moderate versus severe dengue.
DENV1-4 geometric mean titer (GMT) | Enrollment to day 21
  DENV1-4 GMT overtime will be compared between mild/moderate and severe dengue groups. These will also be correlated with disease outcome and GMT at convalescence.
Peak dengue virus enhancing titer | Enrollment to day 21
  Peak dengue virus enhancing titer overtime will be compared between mild/moderate and severe dengue groups. These will also be correlated with disease outcome and GMT at convalescence.
Mean fluorescence intensity of specific lymphocyte populations among groups | Enrollment to day 3
  Mean fluorescence intensity of specific lymphocyte populations will be compared mild/moderate versus severe dengue and dengue versus sepsis.
Number of differentially expressed genes among groups | Enrollment to day 3
  The number of differentially expressed genes will be compared between mild/moderate and severe dengue and dengue versus sepsis based on thresholds for statistical significance (e.g., adjusted p-value < 0.05) and magnitude of change (e.g., absolute log2 fold change > 1).

CONTACTS AND LOCATIONS:
Overall Officials: Tineke Cantaert, PhD, Principal Investigator — Institut Pasteur du Cambodge
Locations (3):
- Cambodia (3):
  - Kampong Speu District Referral Hospital, Kampong Speu
  - International Center of Excellence in Research Cambodia, Phnom Penh
  - Preah Kossamak Hospital, Phnom Penh